CLINICAL TRIAL: NCT06686693
Title: Intravenous Iron Prophylaxis for Rapid High Altitude Insertions
Brief Title: Intravenous Iron Effects on Performance at High Altitude
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Roy Salgado, Principal Investigator, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-24HC (M-10949); 000000 (Other Grant/Funding Number: MRDC)
Record Dates: First submitted 2024-10-31; First posted 2024-11-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: This is a double-blind, parallel research study design where one group will receive iron or placebo intravenously.
Who Masked: Participant, Investigator
Masking Description: Participants and Investigator will be blinded to who receives iron or placebo. A investigator not participating in data collection is responsible for randomly assigning participants to the intervention. The medical care providers will be unblinded to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Experimental): Placebo - saline
  Interventions: Other: Placebo
- Intravenous iron (Experimental): Iron - Injectafer 15 mg/kg up to 1000 mg
  Interventions: Drug: Injectafer

INTERVENTIONS:
Drug: Injectafer — Injectafer - 15 mg/kg up to 1000 mg
  Arms: Intravenous iron
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To compare the effects of IV iron versus placebo (saline) injection on arterial oxygen saturation, submaximal exercise responses, and 2-mile treadmill time-trial performance during acute exposure to hypobaric hypoxia (430 mmHg, simulating ~4800m) assessed 1 and 14 days after treatment.

Primary Hypothesis 1: IV iron treatment will improve arterial oxygen saturation at rest and during exercise in acute hypobaric hypoxia and this effect will persist for 2 weeks

Primary Hypothesis 2) IV iron treatment will improve 2-mile treadmill time trial performance in acute hypobaric hypoxia and this effect will persist for 2 weeks

DETAILED DESCRIPTION:
This study will use a double-blind randomized study design in which one group will receive iron (n = 12; Injectafer, 15 mg/kg up to 1000 mg) and the other a placebo (n = 12; saline). Twenty-four participants will complete seven study visits: Visit 1: Orientation visit consisting of dual-energy X-ray absorptiometry scan (DEXA), pulmonary function test, assessment of peak aerobic capacity (VO2peak); Visits 2-3: familiarization consisting of exercise battery (20 minutes of walking followed by 2 mile treadmill time trial); Visits 4, 6-7: high altitude trial (4,800 m) in which skin blood flow during rest will be measured, ventilation at sea level and altitude will be assessed, collection of sea level and altitude arterialized capillary and venous blood will be collected, and the exercise battery. Visit 5: participants will receive the iron or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, age 18-40 years

  * BMI 18.5-30 kg/m2
  * In good health as determined by the Office of Medical Support & Oversight (OMSO) General Medical Clearance
  * Passed his/her most recent Army Combat Fitness Test (ACFT) (Military Volunteers Only) or exercises at least 2 times per week and able to complete two mile run in ≤ 21 minutes (Civilian Volunteers)
  * Willing to not exercise, or drink alcoholic/caffeinated beverages 24 hours prior to each testing session
  * Willing to not perform any strenuous exercise 36 hours prior to each testing session

Exclusion Criteria:

* Women who are pregnant or planning to become pregnant during the study

  * Taking prescription medication, or over-the-counter medications other than contraceptives, unless approved by OMSO & PI
  * Taking dietary supplements unless approved by OMSO & PI
  * Born at altitudes greater than 2,100 m (7,000 ft)
  * Living in areas that are more than 1,200 m (4,000 ft) or have traveled to areas that are more than 1,200 m for five days or more within the last 2 months
  * Prior diagnosis of High Altitude Pulmonary Edema (HAPE) or High Altitude Cerebral Edema (HACE)
  * Musculoskeletal injuries that compromise the ability to walk/run on a treadmill
  * Presence of abnormal blood chemicals (hemoglobin S or Sickle Cell Trait)
  * Hemoglobin concentration: men: Hb <13.5 g/dL or Hb >17.7 g/dL; women Hb <12.5 g/dL or Hb >15.9 g/dL
  * Ferritin < 50 ng/mL or greater than 150 ng/mL
  * Any history of malignancy
  * Personal or family history of blood clots
  * History of thromboembolic disease, hypertension, and known risk factors of cardiovascular disease
  * Blood donation within 8 weeks of beginning the study
  * History of seizures
  * History of inflammatory bowel disease
  * Any recent (within 4-6 weeks) and or expected history of prolonged periods of immobility or limited activity (including recent or upcoming surgery)
  * Abnormal PT/PTT test or problems with blood clotting
  * Any nicotine or recreational drug use (unless quit > 1 month prior to study orientation)
  * Presence of respiratory tract infections (< 1 month prior)
  * Experience recent cold, coughs, or sinus infections (< 2 weeks prior)
  * Allergy to skin adhesive
  * Evidence of apnea or sleeping disorder
  * Present condition of alcoholism, use of anabolic steroids, other substance abuse issues
  * Body mass <50 kg (110.5 lbs)
  * History of hyperparathyroidism
  * History of vitamin D deficiency
  * History of systemic inflammatory disease (rheumatoid arthritis, lupus erythematosus)
  * Any drug allergies
  * History of hypersensitivity reaction
  * History of asthma
  * History of kidney or liver disease
  * Any previous intravenous iron injection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
2 mile treadmill time trial performance | Baseline at sea level, pre intervention at altitude, one week post intervention at altitude, and two weeks post intervention at altitude.
  Time to complete self-paced 2 miles treadmill time trial (min:sec)

SECONDARY OUTCOMES:
Ventilation rate | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Ventilation rate will be assessed using a pneumotachometer (l/min).
Percent body fat | Will be assessed once at the beginning of the study.
  Percent body fat will be assessed using Dual Energy X-ray Absorptiometry (%body fat).
Oxygen Saturation | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Oxygen saturation will be assessed using a finger pulse oximeter (%).
Hematocrit | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Hematocrit will be assessed using manual hematocrit method (%).
Ferritin | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Ferritin will be assessed using an ELISA (ng/ml).
C-reactive protein | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  C-reactive protein will be assessed using an ELISA (mg/L).
Soluble transferrin | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Soluble transferrin will be assessed using an ELISA (mg/L).
Arterialized capillary PO2 | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Arterialized capillary PO2 will be assessed using a blood gas analyzer (mmHg).
Arterialized capillary PCO2 | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Arterialized capillary PCO2 will be assessed using a blood gas analyzer (mmHg).
Arterialized capillary pH | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Arterialized capillary pH will be assessed using a blood gas analyzer.
Skin Blood flow | Pre intervention at sea level and altitude, one week post intervention at sea level and altitude, and two weeks post intervention at sea level and altitude.
  Skin blood flow will be assessed via laser doppler (arbitrary units).
VO2peak | Will be assessed once on day 1.
  Peak aerobic capacity will be assessed using a metabolic cart (ml/kg/min and or l/min).
Pulmonary function test | Will be assessed once on day 1.
  Pulmonary function test will be performed to determine forced vital capacity (FVC; L) using a metabolic cart.
Pulmonary function test | Will be measured once on day 1.
  Pulmonary function test will be performed to determine forced expired volume in one second (FEV1; L) using a metabolic cart.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Salgado, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States